CLINICAL TRIAL: NCT01000272
Title: Pulmonary Inflammation in Children With Inflammatory Bowel Disease as Expressed by the Fraction of Exhaled Nitric Oxide Levels and Spirometry
Brief Title: Respiratory Tract Inflammation in Children With Inflammatory Bowel Disease (IBD)
Status: Completed | Type: Observational
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Sponsor
Other Study IDs: TASMC-09-YS-439-CTIL
Record Dates: First submitted 2009-10-20; First posted 2009-10-23 (Estimated); Last update posted 2014-06-26 (Estimated); Status verified 2009-10

CONDITIONS: Inflammatory Bowel Disease
MeSH Terms: conditions — Inflammatory Bowel Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to determine whether inflammatory bowel disease in children involve the respiratory tract as expressed by increased levels of the Fraction of exhaled Nitric Oxide (FeNO) and spirometry.

DETAILED DESCRIPTION:
Inflammatory bowel disease, Crohn's disease (CD) and Ulcerative colitis (UC) are chronic inflammatory diseases with remissions and exacerbations. CD and UC are associated with a variety of systemic (extra-intestinal) manifestations. In some studies, clinical and subclinical pulmonary abnormalities are described in active IBD as well as in the stable situation.

Nitric oxide (NO) is an important mediator of inflammation in several pathological conditions.Patients with lung diseases, like asthma, have higher levels of the Fraction of exhaled Nitric Oxide (FeNO) in active disease in comparison with healthy volunteers. One study in adult IBD patients showed increase in FeNO levels in those patients, with positive correlation with the disease activity and negative correlation between the disease activity and pulmonary functions.

We hypothesised that respiratory tract inflammation as expressed by FeNO and spirometry in pediatric IBD patients will correlate to the activity of the primary disease.

Methods: FeNO levels and spirometry will be assess for 40 patients with CD or UC (age 4-18 years) during remissions and exacerbations, calculated by the Pediatrics Crohn's Disease Activity Index (PCDAI) and the Pediatrics Ulcerative Colitis Activity Index (PUCAI), respectively.

Two aged matched groups, the first of healthy children and the second of chronic abdominal pain will serve a controls.

ELIGIBILITY:
Inclusion Criteria:

1. 4-18 years old children diagnosed with IBD:

   * Histological diagnosis of Crohn's disease
   * Histological diagnosis of Ulcerative colitis
2. Negative stool cultures

Exclusion Criteria:

1. Respiratory tract infection during the 6 weeks prior to enrollment
2. Diagnosis of asthma
3. Current treatment with steroids
4. Smoking

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: pediatric patients with IBD addmited to the pediatric ward due to exacerbations and children with IBD who come for routine visit to the pediatric gastroenterology clinic at the "DANA" Hospital for Childrens, at the Sourasky Medical Center, Tel-Aviv
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2009-12; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Fraction of exhaled Nitric Oxide (FeNO) | 1 year

SECONDARY OUTCOMES:
Spirometry | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Yakov Sivan, Associate Professor, Principal Investigator — Tel Aviv Medical Center
Locations (1):
- "DANA" childrens hospitall, Tel Aviv, Israel